CLINICAL TRIAL: NCT05250167
Title: Skeletal Muscle Oxygenation in Patients With Chronic Kidney Disease Stage 2, 3 and 4
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Marieta Theodorakopoulou, PhD Candidate, Aristotle University Of Thessaloniki
Other Study IDs: ΔΔ4871
Record Dates: First submitted 2022-02-06; First posted 2022-02-22 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Diseases
Keywords: chronic kidney disease; NIRS; muscle oxygenation; cerebral oxygenation; microvascular function
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- CKD patients stage 2
- CKD patients stage 3a
- CKD patients stage 3b
- CKD patients stage 4
- Controls without CKD

SUMMARY:
Endothelial dysfunction occurs early in chronic kidney disease (CKD) and is associated with target organ damage, progression of renal injury, cardiovascular events, and mortality. Near-infrared spectroscopy (NIRS) is a relevant new, noninvasive method that assesses local tissue oxygenation and can provide valuable information about local oxygen consumption and blood flow. Using postocclusion reactive hyperemia, NIRS technology provides valuable information on skeletal muscle's oxidative capacity, microvascular function, and muscle oxygenation at rest and during exercise. With regard to cerebral oxygenation, NIRS noninvasively monitors alterations and assesses relative changes from baseline for oxygenated, deoxygenated, and total hemoglobin. Due to its ability to assess microvascular function, NIRS has been applied in various populations with impaired microvascular function, including patients with hypertension, diabetes, CAD, and end-stage kidney disease. However, there is no study up to date assessing muscle oxygenation and microvascular function measured via NIRS in patients with different stages of CKD. Hence, this study aims to examine possible differences in muscle and oxygenation at rest, exercise, and during an occlusion-reperfusion maneuver in CKD stages 2-4 with NIRS. In addition, this is the first study examining potential associations between micro-, macrovascular dysfunction and potentially impaired muscle and cerebral oxygenation in CKD patients.

DETAILED DESCRIPTION:
This is a cross-sectional study performed in the Department of Nephrology, Hippokration Hospital, Thessaloniki, Greece. For the purposes of this study, consecutive CKD patients stage 2-4 regularly followed in outpatient clinics of the Department of Nephrology, and fulfilling the inclusion/exclusion criteria, as well as controls without CKD, were invited to participate. All included patients signed a written informed consent form. The study protocol was approved by the Ethics Committee of the School of Medicine, Aristotle University of Thessaloniki. All procedures and evaluations are performed according to the Declaration of Helsinki 2013 Amendment.

Baseline evaluation includes the recording of demographics, anthropometric characteristics, CKD cause, comorbidities, concomitant medications, and a detailed physical examination. The Mini-Mental State Exam (MMSE) is used for the assessment of cognitive function; physical activity status is evaluated by the International Physical Activity Questionnaire. Study participants are advised to refrain from food, caffeine, alcohol, or tobacco for 12 h and received any standard medication before their morning appointment in the research laboratory to perform the assessments described below. BP measurements are performed thrice after 10 min of rest, in the sitting position, at the level of the brachial artery, with a validated oscillometric device [Omron M3 Intellisense (Omron Healthcare, Kyoto, Japan)] and a cuff of appropriate size, according to current guidelines. Afterwards, venous blood samples are collected for routine laboratory parameters. Office arterial stiffness and arterial wave parameters are measured with applanation tonometry using the Sphygmocor device (AtCor, Sydney, Australia). The common carotid intima-media thickness (cIMT) is measured with a 2D ultrasound device (GE Healthcare Ultrasound, Vivid S5, 8L-RS probe, USA) in the CCA between the middle and inner surface of the right and left artery wall, which is represented by a dense double-line pattern. Next, the participant is connected to the experimental apparatus for assessment of muscle and cerebral oxygenation via NIRS (Artinis, The Netherlands). The NIRS device is placed: a) on the forearm of the dominant limb for non-invasive monitoring of skeletal muscle oxygenation (absolute values and relative changes from baseline for oxygenated, deoxygenated, and total hemoglobin as well as tissue saturation index (TSI), as an absolute parameter for muscle oxygenation), and b) over the prefrontal cortex (contra-laterally of the dominant arm), 2 cm beside the midline and about 3 cm above the supraorbital ridge for assessing cerebral oxygenation. In brief, after calibration, with the participant in the seated position, baseline values are obtained, and a 5-minute arterial occlusion is performed. The cuff is rapidly inflated to suprasystolic levels (ie, 250 mm Hg), to obstruct blood flow to forearm muscles and measure the maximal capacity for oxygen extraction by skeletal muscles. Stable blood flow/volume is verified by total hemoglobin. The cuff is then rapidly deflated, and reoxygenation responses are recorded. After a subsequent 10-minute rest, the participant's maximal voluntary contraction (MVC) is assessed, using a digital dynamometer (K-Force, K-invent), followed by a 3-minute submaximal handgrip exercise test (set of 30 s exercise at 35% MVC with 3 s rest). The participant has visual feedback to maintain the force output to the predetermined MVC percentage. At the completion of the exercise protocol, the Rate of Perceived Exertion (RPE) is assessed using the the Borg scale. Continuous beat-by-beat SBP/DBP are recorded by photo-plethysmography (Finometer pro, Finapres Medical Systems, Amsterdam, The Netherlands) throughout the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Patients with CKD stage 2, 3a, 3b, 4 (CKD-EPI eGFR: <90 and ≥30mL / min / 1.73m2) and controls without CKD
* Provision of informed written signed consent prior to study entry

Exclusion Criteria:

* Kidney transplant recipients
* Myocardial infarction or unstable angina episode within the past 3 months, or congestive heart failure class III-IV according to New York Heart Association criteria
* Patients with history of stroke, dementia or other severe neurologic disorders (e.g. Parkinson's disease, multiple sclerosis, etc)
* Patients with severe mental disorders
* History of drug or alcohol abuse
* Patients with muscle disorders
* Active malignant disease or other comorbidity with poor prognosis
* Active infection or relevant inter-current illness
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study includes patients with CKD stage 2, 3a, 3b and 4 (CKD-EPI eGFR: <90 και ≥30mL/min/1.73m2) and controls without CKD.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in skeletal muscle oxygen saturation (TSI%) at rest. | Baseline

SECONDARY OUTCOMES:
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle TSI slope during occlusion | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle TSI magnitude during occlusion | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle oxygen consumption during occlusion | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in the hyperemia range (calculated as the difference between maximal TSI during reperfusion and rest TSI) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle TSI slope during reperfusion | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle TSI magnitude during reperfusion | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle oxygenation during a 3-min handgrip exercise (35% of maximal voluntary capacity) (TSI change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle oxygenation during a 3-min handgrip exercise (35% of maximal voluntary capacity) (O2Hb change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle oxygenation during a 3-min handgrip exercise (35% of maximal voluntary capacity) (HHb change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in muscle total blood volume during a 3-min handgrip exercise (35% of maximal voluntary capacity) (tHb change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in cerebral oxygenation at rest (TSI) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in cerebral oxygenation during a 3-min handgrip exercise (35% of maximal voluntary capacity) (TSI change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in cerebral oxygenation during a 3-min handgrip exercise (35% of maximal voluntary capacity) (O2Hb change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in cerebral oxygenation during a 3-min handgrip exercise (35% of maximal voluntary capacity) (HHb change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in cerebral total blood volume during a 3-min handgrip exercise (35% of maximal voluntary capacity) (tHb change from baseline) | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in office pulse wave velocity. | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in office augmentation pressure and augmentation index. | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in office central systolic and diastolic blood pressure | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in office brachial systolic and diastolic blood pressure | Baseline
Differences between CKD stages (stage 2, 3a, 3b and 4) and controls in carotid intima-media thickness | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nephrology, Hippokration Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Theodorakopoulou MP, Schoina M, Sarafidis P. Assessment of Endothelial and Microvascular Function in CKD: Older and Newer Techniques, Associated Risk Factors, and Relations with Outcomes. Am J Nephrol. 2020;51(12):931-949. doi: 10.1159/000512263. Epub 2020 Dec 11. PMID 33311014
- [Background] Dipla K, Triantafyllou A, Koletsos N, Papadopoulos S, Sachpekidis V, Vrabas IS, Gkaliagkousi E, Zafeiridis A, Douma S. Impaired Muscle Oxygenation and Elevated Exercise Blood Pressure in Hypertensive Patients: Links With Vascular Stiffness. Hypertension. 2017 Aug;70(2):444-451. doi: 10.1161/HYPERTENSIONAHA.117.09558. Epub 2017 Jun 12. PMID 28607132
- [Background] Moody WE, Edwards NC, Madhani M, Chue CD, Steeds RP, Ferro CJ, Townend JN. Endothelial dysfunction and cardiovascular disease in early-stage chronic kidney disease: cause or association? Atherosclerosis. 2012 Jul;223(1):86-94. doi: 10.1016/j.atherosclerosis.2012.01.043. Epub 2012 Feb 2. PMID 22349087
- [Background] Kintiraki E, Dipla K, Triantafyllou A, Koletsos N, Grigoriadou I, Poulakos P, Sachpekidis V, Vrabas IS, Zafeiridis A, Bili E, Douma S, Goulis DG. Blunted cerebral oxygenation during exercise in women with gestational diabetes mellitus: associations with macrovascular function and cardiovascular risk factors. Metabolism. 2018 Jun;83:25-30. doi: 10.1016/j.metabol.2018.01.009. Epub 2018 Feb 2. PMID 29410188